CLINICAL TRIAL: NCT01574365
Title: A Phase 2 Study of RTA 402 in CKD Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of RTA 402 in Chronic Kidney Disease (CKD) Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTA 402-003
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
Keywords: CKD patients with type 2 diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RTA402 (Experimental)
  Interventions: Drug: RTA 402
- RTA402 Low (Experimental)
  Interventions: Drug: RTA 402
- RTA402 Medium-low (Experimental)
  Interventions: Drug: RTA 402
- RTA402 Medium-high (Experimental)
  Interventions: Drug: RTA 402

INTERVENTIONS:
Drug: RTA 402

SUMMARY:
A Phase 2 study of RTA 402 in Chronic kidney disease (CKD) patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of RTA 402 in patients with type 2 diabetes mellitus.

To evaluate the safety and tolerability of RTA 402.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with type 2 diabetes mellitus
* Patients whose eGFR levels are eligible for this study
* Patients being treated with stable dose of ACE inhibitors and/or ARB etc.

Exclusion Criteria:

* Patients with Type 1 diabetes
* Patients with known non-diabetic renal disease
* Patients with a history of renal transplantation
* Patients with mean SBP > 160 mmHg or mean DBP > 90 mmHg
* Patients with HbA1C > 10%
* Patients with cardiovascular disease specified in the study protocol etc.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Efficacy:Changes in eGFR | Up to 16 weeks
  Changes in eGFR from baseline to the study week 12 or to the time of treatment discontinuation.
Adverse event collection and assessment | Up to 16 weeks
  Adverse Event collection and assessment will be done for all treated subjects.

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | Baseline, week 4, 8 and 12.
  Relationship between the study drug dose and the trough concentration of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Toride, Ibaraki, Japan